CLINICAL TRIAL: NCT07262476
Title: A Phase III, Multicenter, Open-Label Extension Study to Evaluate the Efficacy and Safety of MHB018A Injection in Subjects With Thyroid Eye Disease
Brief Title: Open-Label Extension Study of MHB018A in Subjects With Thyroid Eye Disease
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Minghui Pharmaceutical (Hangzhou) Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MHB018A-P-303
Record Dates: First submitted 2025-11-20; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Thyroid Eye Disease (TED)
MeSH Terms: conditions — Graves Ophthalmopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MHB018A Injection (Experimental): Subcutaneous injections of MHB018A injection, 450mg once every 4 weeks (q4w).
  Interventions: Drug: MHB018A injection

INTERVENTIONS:
Drug: MHB018A injection — MHB018A 450mg for subcutaneous injection once every 4 weeks (Q4W)

SUMMARY:
This is a multicenter, open-label extension (OLE) study of MHB018A in subjects with moderate-to-severe TED.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the improvement in proptosis from baseline (defined as the most recent measurement prior to the first dose in this study) following treatment with MHB018A Injection in subjects with active or chronic TED who previously received placebo in either the MHB018A-P-301 or MHB018A-P-302 studies, and the safety and tolerability of MHB018A Injection in TED subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily participating in the study and signing the informed consent form;
2. Aged 18-75 years (inclusive), of any gender;
3. Completed the 24-week double-blind treatment period in either the MHB018A-P-301 or MHB018A-P-302 study, and within 28 days after Week 24 visit of the previous study when enrolled in this OLE study (does not apply to subjects who meet the relapse criteria during the safety follow-up period).
4. Proptosis non-responder at Week 24 visit in the double-blind treatment period of either the MHB018A-P-301 or MHB018A-P-302 study (defined as a <2 mm reduction from baseline in the study eye, or a ≥2 mm reduction in the study eye accompanied by a ≥2 mm worsening from baseline in proptosis of the fellow eye), and/or who meet the retreatment criteria for relapse during the safety follow-up period.
5. Does not require immediate surgical ophthalmological intervention, and no corrective surgery/orbital radiotherapy is planned during the study.
6. Diabetic subjects must have well-controlled stable disease.
7. Sufficient bone marrow and organ function.
8. Eligible subjects of childbearing potential (male and female) must agree to use reliable contraceptive methods; female subjects of childbearing potential must have a negative blood pregnancy test within 7 days before the first use of the study drug and must not be breastfeeding.
9. Subject is willing and able to comply with the prescribed treatment protocol and evaluations for the duration of the study.

   -

Exclusion Criteria:

1. Decreased best corrected visual acuity due to optic neuropathy as defined by a decrease in vision within the last 6 months of two lines of Snellen chart, new visual field defect or color defect secondary to optic nerve involvement.
2. Corneal decompensation unresponsive to medical management.
3. Free thyroxine (FT4) and free triiodothyronine (FT3) levels <50% above or below the normal reference range at screening.
4. Received any treatment for TED, intravenous corticosteroids, immunosuppressive agents, investigational drug from the last visit of the MHB018A-P-301 or MHB018A-P-302 trial until participation in this study.
5. Identified pre-existing ophthalmic disease that would preclude study participation or complicate interpretation of the study results.
6. Acute cardiovascular disease history or treatment within 6 months before the first dose from the last visit of the MHB018A-P-301 or MHB018A-P-302 trial until participation in this study.
7. Presence of poorly controlled hypertension with systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg; Renal artery stenosis.
8. Pregnant or lactating women.
9. Tinnitus or other hearing impairment.
10. Poor compliance or severe systemic disease history or other reasons that make the subject unsuitable for participation in this clinical study.

    -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Proptosis Responder Rate at Week 24 | Week 24
  The proptosis response rate at Week 24 in the study eye for subjects with active or chronic TED who received MHB018A placebo in either the MHB018A-P-301 or MHB018A-P-302 studies: the proportion of subjects achieving a reduction of ≥2 mm in proptosis from baseline (defined as the most recent measurement prior to the first dose in this study) in the study eye, without deterioration in the other eye (defined as an increase in proptosis of ≥2 mm).

SECONDARY OUTCOMES:
TED relapse rate | From baseline up to Week 24
  TED relapse rate from treatment discontinuation to relapse (for subjects with active or chronic TED who previously received and completed 24 weeks of MHB018A Injection treatment in either the MHB018A-P-301 or MHB018A-P-302 study, meet the disease relapse enrollment criteria for this study during the safety follow-up period, and receive retreatment with MHB018A Injection)
TED relapse time | Up to Week 24 and at end-of-trial (EOT) visit
  TED relapse time from treatment discontinuation to relapse (for subjects with active or chronic TED who previously received and completed 24 weeks of MHB018A Injection treatment in either the MHB018A-P-301 or MHB018A-P-302 study, meet the disease relapse enrollment criteria for this study during the safety follow-up period, and receive retreatment with MHB018A Injection)
Overall response rate | Week 24
  The percentage of subjects with ≥2-points in Clinical Activity Score (CAS) reduction and ≥2 mm reduction in proptosis from baseline, provided there is no corresponding deterioration (≥2-points/mm increase) in CAS or proptosis in the fellow eye.
Change in proptosis | Baseline, up to Week 24
  Change from baseline in proptosis in the study eye as measured by exophthalmometer at Week 24
Percentage of subjects with CAS of 0 or 1 | Week 24
  The percentage of subjects with a CAS of 0 or 1 in the study eye/target eye.
Change in CAS | Week 24
  The mean change from baseline to Week 24 in the CAS in the study eye/target eye.
Diplopia response rate | Week 24
  The percentage of subjects with a reduction in diplopia severity by ≥1 grade.
Change in Quality of Life (GO-QOL) Scores | Up tp Week 24
  The mean change in scores from the Graves' Ophthalmopathy Quality of Life questionnaire compared to baseline. The GO-QoL is a self-filled questionnaire containing 16 items. The raw scores for items 1-8 and items 9-16 are summed separately, each yielding a total raw score ranging from 8 to 24. Each raw score is then transformed into a 0-100 scale using the following formula: Total Score = (Raw Score - 8) ÷ 16 × 100. Higher scores indicate better quality of life.
Pharmacokinetic Parameter Trough Concentration for MHB018A | Up tp Week 24
  Trough concentration (Ctrough) will be assessed using non-compartmental methods in participants randomized to the MHB018A group.
Incidence of Adverse Events (AEs) During Treatment | Up to Week 24 and at end-of-trial (EOT) visit
  Including Treatment-Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), and AEs leading to early study withdrawal, along with laboratory tests, 12-lead ECGs, vital signs, and physical examinations.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ninth People's Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No